CLINICAL TRIAL: NCT03260231
Title: Effects of Dietary Milled Seed Mix in Patients With Non-Hodgkin Lymphoma
Brief Title: Dietary Milled Seed Mix in Patients With Non-Hodgkin Lymphoma
Acronym: Lymphoseed
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Belgrade (Other)
Responsible Party: Principal Investigator, Vesna Vucic, Professor of Research, University of Belgrade
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 145/1
Record Dates: First submitted 2017-08-11; First posted 2017-08-24 (Actual); Last update posted 2020-03-20 (Actual); Status verified 2020-03

CONDITIONS: Non-hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin

STUDY DESIGN:
Intervention Model Description: This study is a parallel, randomized, single blind, controlled, 5-months nutritional intervention, investigating health effects of dietary intake of milled mix of flax/sesame pumpkin seeds in sour milk, in patients with NHL undergoing chemotherapy.
  At the beginning of the study, all patients received nutritional counselling, where half of the study subjects are randomly assigned to a treatment arm with milled seed mix consumption, or control arm without seed mix. Treatment arm is provided with 450g of milled seed mix and instructed to consume 30g of the mix daily (18g flax seed, 6g pumpkin seeds, and 6 g sesame) in 180 mL of sour milk. Control arm is instructed to consume180 mL of sour milk.
Who Masked: Care Provider, Investigator
Masking Description: Single blind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Active Comparator): Dietary Supplement: Milled Seed Mix Intervention arm includes milled mix of flax, sesame and pumpkin seeds (18/6/6 g) in sour milk taken as dietary replacement meal during the day, and between lunch and dinner. Seeds are provided with the same producer at the Belgrade market.
  Interventions: Dietary Supplement: Milled seed mix
- Control group (No Intervention): No supplement Control arm includes nutritional counseling with a similar dietary regime as for the intervention arm, but without milled seed mix. patients were instructed to avoid plant seeds during the study.

INTERVENTIONS:
Dietary Supplement: Milled seed mix — Dietary intervention with or without seed mix
  Arms: Intervention group

SUMMARY:
Recent literature data suggest beneficial effects of dietary fats in patients with cancers, in particular polyunsaturated fatty acids (PUFAs). Milled mix of flax, sesame and pumpkin seeds provides a high amount of PUFAs and a desirable n-6/n-3 PUFAs ratio.

DETAILED DESCRIPTION:
Cancers are characterized by inflammation and alternations in lipid and fatty acid metabolism. Patients with non-Hodgkin lymphoma have impaired fatty acid profiles, low level of PUFAs, and high n-6/n-3 PUFAs ratio. Moreover, these changes are related to clinical outcome.

Flax seeds, sesame and pumpkin seeds are rich sources of PUFAs. Dietary intake of milled mix of these seeds has been shown to decrease inflammation and improve PUFAs status in patients on hemodialysis and to decrease breast cancer risk.

The study design is single-blind, controlled, randomized nutritional intervention. The participants are randomly assigned into intervention and control group before starting chemotherapy. All patients receive nutritional counseling to achieve a daily energy and protein intake according to recommended dietary allowances, with (intervention) or without (control) of milled seed mix.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed Non-Hodgkin lymphoma
* Patients able to understand requirements of the study and provide written informed consent

Exclusion Criteria:

* Previous radio- or chemotherapy
* Other serious chronic diseases
* Statin therapy
* Presence of allergy on any seeds
* Use of fat-based dietary supplements (such as fish oil, evening primrose oil etc) 3 months prior to study

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-05-12 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in disease status | Baseline, 5 months, 1 year
  Remission, stable disease or progression
Change in quality of life questionnaire scores | Baseline, 5 months, 1 year
  Assessed by standardized questionnaires

SECONDARY OUTCOMES:
Changes in body weight | Baseline, 5 months, 1 year
  Changes in body weight measured by bio-impedance analyzer, from baseline to endpoint
Changes in leukocyte count | Baseline, 5 months, 1 year
  Measures of leukocyte count
Changes in lipid profiles | Baseline, 5 months, 1 year
  Changes in lipid profiles (cholesterol, HDL, LDL and triglycerides) from baseline to endpoint
Changes in plasma fatty acids | Baseline, 5 months, 1 year
  Changes in plasma fatty acids profiles from baseline to endpoint
Changes in CRP | Baseline, 5 months, 1 year
  Changes in CRP from baseline to endpoint
Changes in interleukin (IL)-6 | Baseline, 5 months, 1 year
  Changes in interleukin (IL)-6 from baseline to endpoint
Changes in parameters of oxidative stress | Baseline, 5 months
  Measures of activities of the following enzymes: SOD, catalase, glutathion peroxidase and glutation reductase

CONTACTS AND LOCATIONS:
Overall Officials: Vesna Vucic, PhD, Principal Investigator — Institute for medical research
Locations (1):
- Center of Research Excellence in Nutrition and Metabolism, Institute for Medical Research, University of Belgrade, Belgrade, Serbia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cvetkovic Z, Milosevic M, Cvetkovic B, Masnikosa R, Arsic A, Petrovic S, Vucic V. Plasma phospholipid changes are associated with response to chemotherapy in non-Hodgkin lymphoma patients. Leuk Res. 2017 Mar;54:39-46. doi: 10.1016/j.leukres.2017.01.004. Epub 2017 Jan 5. PMID 28107691
- [Background] Cvetkovic Z, Vucic V, Cvetkovic B, Petrovic M, Ristic-Medic D, Tepsic J, Glibetic M. Abnormal fatty acid distribution of the serum phospholipids of patients with non-Hodgkin lymphoma. Ann Hematol. 2010 Aug;89(8):775-82. doi: 10.1007/s00277-010-0904-6. Epub 2010 Feb 3. PMID 20127484
- [Background] Ristic-Medic D, Perunicic-Pekovic G, Rasic-Milutinovic Z, Takic M, Popovic T, Arsic A, Glibetic M. Effects of dietary milled seed mixture on fatty acid status and inflammatory markers in patients on hemodialysis. ScientificWorldJournal. 2014 Jan 22;2014:563576. doi: 10.1155/2014/563576. eCollection 2014. PMID 24578648